CLINICAL TRIAL: NCT01411293
Title: Vasoprotective Activities of Low-Fat Milk in Individuals With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Richard Bruno, Principal Investigator, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H11-124
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Disease; Metabolic Syndrome; Obesity
Keywords: cardiovascular disease; oxidative stress; dairy consumption; metabolic syndrome; obesity; endothelial function
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome; Obesity | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Fat Dairy (Experimental): Participants will ingest 2 cups of low-fat milk on 1 occasion prior to measure postprandial changes in vascular function
  Interventions: Other: Low-Fat Milk
- Rice Milk (Active Comparator): Participants will ingest 2 cups of rice milk on 1 ocassion prior to measuring postprandial vascular function
  Interventions: Other: Rice Milk

INTERVENTIONS:
Other: Low-Fat Milk — Participants will ingest 2 cups of low-fat milk on 1 occasion.
  Arms: Low-Fat Dairy
Other: Rice Milk — Participants will ingest 2 cups of rice milk on 1 occasion.
  Arms: Rice Milk

SUMMARY:
The purpose of this study is to define whether the acute consumption of low-fat milk protects against postprandial vascular endothelial dysfunction by reducing oxidative stress responses that limit nitric oxide bioavailability to the vascular endothelium. The investigators hypothesis is that the consumption of low-fat milk will improve postprandial vascular endothelial function in an oxidative stress-dependent manner that allows greater nitric oxide (NO) bioavailability. The objectives of this study are to 1) examine improvements in postprandial vascular endothelial function in response to low-fat milk ingestion, 2) define low-fat milk-mediated improvements in circulating biomarkers of redox status, and 3) define the mechanism by which low-fat milk improves NO bioavailability. Collectively, the successful completion of these studies is expected to define NO mediated activities of low-fat milk that protect against vascular endothelial dysfunction in individuals at high risk for developing CVD.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the United States, accounting for ~830,000 deaths annually. Oxidative stress and inflammatory responses are fundamental mechanisms leading to vascular endothelial dysfunction because of their role in reducing nitric oxide (NO) bioavailability. Greater intakes of dairy foods have been associated with a lower incidence of CVD-related morbidity. Although the mechanisms by which dairy protects against CVD remain unclear, epidemiological and experimental evidence suggest that the concerted actions of bioactive milk-derived peptides and micronutrients may protect against hypertension and future CVD risk by improving vascular endothelial function. Therefore, the objective of this study is to define the mechanisms by which the acute consumption of low-fat milk protects against postprandial vascular endothelial dysfunction by reducing oxidative stress responses that limit NO bioavailability to the vascular endothelium. In this study, participants having the metabolic syndrome will ingest low-fat milk or rice milk on a single occasion. Then, vascular function and biomarkers of oxidative stress and NO metabolism will be monitored at 30 min intervals throughout a 180 min postprandial period. Collectively, these studies will help identify how postprandial vascular function is regulated in individuals at high-risk for CVD, and whether low-fat dairy consumption can be used as a strategy to better improve vascular function.

ELIGIBILITY:
Inclusion Criteria:

* specific criteria of the metabolic syndrome (waist circumference (102-137 or 88-123 cm for men and women, respectively), fasting triglycerides 150-300 mg/dL, and fasting glucose (110-180 mg/dL)
* BMI: >30 kg/m2,
* non-dietary supplement users for >2-mo
* no use of any prescription or over-the-counter medications known to affect vasodilatory responses
* no known history of vascular disease
* nonsmokers
* resting blood pressure <140 mmHg
* not taking any medications that control hypertension

Exclusion Criteria:

* lactose-intolerant
* excessive alcohol consumption (>3 drinks/d or >10 drinks/wk)
* >7 h/wk of aerobic activity
* use of medications known to affect carbohydrate or lipid/lipoprotein metabolism
* regular use of any anti-inflammatory medications (e.g. aspirin, non-steroidal anti-inflammatory drugs) or over-the-counter aids (e.g. fish oils)
* women who are pregnant, lactating, and have initiated or changed birth control in the past 3-mo

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
endothelial function | 3 hours
  Brachial artery flow-mediated dilation will be assessed at 30 min intervals during a 3 hour postprandial period

SECONDARY OUTCOMES:
Biomarkers of oxidative stress and nitric oxide metabolism | 3 hours
  At 30 min intervals throughout a 3 hour postprandial period, biomarkers of oxidative stress (glutathione, malondialdehyde, nitrotyrosine, and antioxidants) as well as nitric oxide metabolism (arginine, asymmetric dimethylarginine, and nitric oxide metabolites) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Bruno, PhD, RD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Result] Ballard KD, Mah E, Guo Y, Pei R, Volek JS, Bruno RS. Low-fat milk ingestion prevents postprandial hyperglycemia-mediated impairments in vascular endothelial function in obese individuals with metabolic syndrome. J Nutr. 2013 Oct;143(10):1602-10. doi: 10.3945/jn.113.179465. Epub 2013 Aug 21. PMID 23966328